CLINICAL TRIAL: NCT05087706
Title: Exploratory Study of Molecular Profile-Associated Evidence Guided Precision Therapy for Salivary Gland Cancer
Brief Title: Exploratory Study of Molecular Profile-Associated Evidence Guided Precision Therapy for Salivary Gland Cancer（MAPS）
Acronym: MAPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021HNRT03
Record Dates: First submitted 2021-09-22; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Salivary Gland Neoplasms
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — pyrotinib; bicalutamide; Leuprolide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Locally advanced patients with molecular-guided therapy: Locally advanced patient will be assigned to molecularly-guided therapy based on genomic profile.
  Interventions: Drug: Pyrotinib; Drug: Bicalutamide; Drug: Leuprorelin
- Advanced patients with molecular-guided therapy: Advanced patient will be assigned to molecularly-guided therapy based on genomic profile.
  Interventions: Drug: Pyrotinib; Drug: Bicalutamide; Drug: Leuprorelin

INTERVENTIONS:
Drug: Pyrotinib — Pyrotinib 400mg qd po
Drug: Bicalutamide — Bicalutamide was administered orally at a daily dose of 50 mg
Drug: Leuprorelin — Leuprorelin acetate was administered subcutaneously at a dose of 3.75 mg every 4 weeks

SUMMARY:
To explore the feasibility, efficacy and safety of determining the treatment regimen based on genomic profiling in patients with locally advanced and advanced salivary gland cancer.

DETAILED DESCRIPTION:
This is a prospective, open-label, non-randomized single-center study to evaluate the feasibility of using molecular profile-based evidence to guide personalized therapy for patients with incurable salivary gland carcinoma patients. Comprehensive Genomic Profiling is performed on tissue with assessment of tumor mutation burden (TMB) status, and additional PD-L1 immunohistochemistry testing. Study Committee or Molecular Tumor Board (MTB) will recommend matched therapy, if available, following analysis of patient genomic profiles. The final treatment administered will be based on the treating physician's choice with MTB advice, patient preference, comorbidity considerations, and available drug access. Access to medication followed real-world practice.

ELIGIBILITY:
Inclusion Criteria for patients with locally advanced gland cancer at high-risk of recurrence must meet all entry criteria for participation in this study:

* Locally advanced salivary gland carcinoma patients with high risk of recurrence confirmed by histology, the main pathological subtypes include:

  * Mucoepidermoid carcinoma
  * Salivary duct carcinoma
  * Non-specific adenocarcinoma
  * Pleomorphic adenocarcinoma, etc.
* Expected survival ≥ 6 months
* Patients with prior standard surgery and post-operative radiotherapy (chemotherapy)
* Adequate function of main organs
* Sufficient tissue samples for gene mutation test
* Signed informed consent

Inclusion Criteria for patients of advanced gland cancer must meet all entry criteria for participation in this study:

* Histologically confirmed recurrent or metastatic salivary gland cancer, the main pathological subtypes include:

  * Mucoepidermoid carcinoma
  * Salivary duct carcinoma
  * Non-specific adenocarcinoma
  * Mastoid secretory carcinoma
  * Pleomorphic adenocarcinoma, etc.
* a measurable lesion according to Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1)
* Expected survival ≥ 6 months
* Adequate function of main organs
* Sufficient tissue samples for gene mutation detection
* Signed informed consent.

Exclusion Criteria for patients with locally advanced disease at high-risk of recurrence who meet any of the exclusion criteria at baseline will be excluded from the study:

* Severe or uncontrolled medical conditions (i.e., uncontrolled diabetes, chronic kidney disease, chronic lung disease or active uncontrolled infection, psychiatric illness/social situations that would, in the opinion of the investigator, confound the analysis of response to study treatment)
* Pregnancy or breastfeeding, or any patient with childbearing potential not using adequate pregnancy prevention

Exclusion Criteria for patients with advanced disease who meet any of the exclusion criteria at baseline will be excluded from the study:

* Primary lesions amenable to local therapy
* Severe or uncontrolled medical conditions (i.e., uncontrolled diabetes, chronic kidney disease, chronic lung disease or active uncontrolled infection, psychiatric illness/social situations that would, in the opinion of the investigator, confound the analysis of response to study treatment).
* Pregnancy or breastfeeding, or any patient with childbearing potential not using adequate pregnancy prevention

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients interviewed at Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Sampling Method: Non-Probability Sample
Enrollment: 182 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2023-03-19 (Estimated); Study Completion 2023-09-19 (Estimated)

PRIMARY OUTCOMES:
Molecular mutation profile of patients with salivary gland cancer | 18 months
  To explore the complete picture of molecular mutations in locally advanced and advanced salivary gland tumors in China
Proportion of patients who receive molecular guided therapy | 18 months
  Proportion of patients who have actionable genomic alterations and receive matched therapy based on genomic profile(s)

SECONDARY OUTCOMES:
Progression-free survival (PFS) in patients | 2 years
  PFS of patients with locally advanced and advanced salivary gland cancer
Objective Response Rate (ORR) | 2 years
  ORR in patients with advanced salivary gland cancer
Overall Survival (OS) | 2 years
  OS of patients with locally advanced and advanced salivary gland cancer
Proportion of patients with actionable genomic alteration | 2 years
  To calculate the proportion of patients with actionable genomic alteration(s)
Treatment-related adverse events (AEs) | 2 years
  The grade of AEs and the number of patients with AEs are assessed by the investigator based on CTCAE v5.0 from the date of enrollment to 90 days after last dose of study treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China